CLINICAL TRIAL: NCT06769230
Title: The Effect of Sensory Motor Training on Postural Stability in Post-menopausal Women With Non-specific Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Khalaf Sayed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005567
Record Dates: First submitted 2025-01-07; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- core strengthening exercise group (Active Comparator): The participants will practice core strengthening exercises (3 sessions/ week) for eight weeks.
  Interventions: Other: Core strengthening exercise
- Core strengthening exercise and sensory motor training group (Experimental): The participants will practice core strengthening exercises and sensory motor training (3 sessions/ week) for eight weeks.
  Interventions: Other: Core strengthening exercise; Other: sensory motor training

INTERVENTIONS:
Other: Core strengthening exercise — The participants will perform warm-up exercises including Cat and Camel, spinal movement (spinal flexion and extension cycles), and stretching exercises for the calf, hamstrings, quadriceps and lower back for about 5 minutes. After that, the women will be asked to perform core stability exercises including abdominal hollowing, bilateral knee raise, supine extension Bridge, straight leg rise from prone and alternate arm and leg raise from quadruped. Each exercise will be repeated for 10 times with 7-8 seconds hold and will be increased by four repetitions each week throughout the interventions. During each repetition for every exercise, the patient will be asked to contract her abdominal muscles and maintain this contraction while maintaining her normal breathing pattern.
Other: sensory motor training — The participants will perform warm-up exercises including neck rotations, arm circles, ankle rotations, trunk rotations, trunk bending and extending for 5-10 mins. After warm up the women performs Bosu ball exercises including Bosu ball one Leg Bridge, Bosu Crunch, Bosu Sit ups, Bosu compressions, Bosu side crunch and Bosu bodyweight squat . Each exercise will be repeated for 6 repetitions in each set. At least 3 sets of each exercise are performed per session. Each exercise will be increased by five repetitions each week throughout the interventions.The total duration of each session is 45 minutes.
  Arms: Core strengthening exercise and sensory motor training group

SUMMARY:
The study will be conducted to determine the effect of sensory-motor training on postural stability in post-menopausal women with non-specific low back pain.

DETAILED DESCRIPTION:
Low back pain (LBP) primarily affects postmenopausal women between the ages of 45-60, and it causes distress on social and economic levels Postmenopausal women with non-specific low back pain (NSLBP) and decreased function often feel anxious and sad, which affects their work, sexual and social lives Neuromuscular rehabilitation techniques addressing sensory deficiencies have emerged in recent years and have received increasing therapeutic attention. These techniques could broadly be summarized as sensorimotor training (SMT) methods aiming at increased proprioceptive input to improve motor response in dynamic environments. This might lead to improved quality of postural control, which in turn may alleviate postural specific musculoskeletal pain.

As it promotes proximal stability and distal mobility, Core muscles Stabilization Exercises (CSE) are becoming a more significant part of the treatments. The use of CSE is promoted as a general physical therapy approach for NSLBP. Overtime, CES have improved, focusing more and more on maintaining spinal stability. Theoretical ideas for the treatment of spinal ailments that aid in reducing pain and enhancing function in patients with LBP significantly support the use of CSE. CSE trains muscle activity patterns without unnecessarily overloading the tissue, enhances aerobic fitness, spinal mobility, muscle strength, motor co-ordination and can help to stabilize the spine at a quite cost affordable price and reduce low back pain.

ELIGIBILITY:
Inclusion Criteria:

* All women suffering from non-specific low back pain for at least 3 months.
* Their ages will be ranged from 50-65 years.
* They will be at least 3 years post menopause.
* Their body mass index (BMI) will be less than 30 kg/m2.

Exclusion Criteria:

* Musculoskeletal injuries.
* Cardiovascular, respiratory or neurological disorders or psychiatric problem.
* Spinal deformity, bone fracture.
* Back surgery experience.
* Hormone replacement therapy and females with cancer.
* Sensory neuropathy and nervous system problems.
* Middle ear or vestibular problems.

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Anterior posterior stability index (APSI) | 8 weeks
  The Biodex Balance System(Model 950-300, Biodex, Inc., Shirley, NY, USA) will be used to assess posture stability including anterior posterior stability index. It offers 12 levels of platform control and provides up to 20⁰ of surface tilt. Before the participant stepped onto the Biodex Balance System, the platform was in the "locked" position. Participants' data and test parameters were inserted. The parameters will be included trial time (20 seconds), number of trials (3 trials), and in between trials rest (10 seconds). Initial and end stability levels will be set from more to less stable (8-1) respectively. Anterior-posterior stability index (APSI) represents fluctuations from the horizontal around the anteroposterior axis. The higher the value, the lower the anterior posterior stability.
Mediolateral stability index (MLSI) | 8 weeks
  The Biodex Balance System(Model 950-300, Biodex, Inc., Shirley, NY, USA) will be used to assess posture stability including mediolateral stability index. It offers 12 levels of platform control and provides up to 20⁰ of surface tilt. Before the participant stepped onto the Biodex Balance System, the platform was in the "locked" position. Participants' data and test parameters were inserted. The parameters will be included trial time (20 seconds), number of trials (3 trials), and in between trials rest (10 seconds). Initial and end stability levels will be set from more to less stable (8-1) respectively. Medio-lateral stability index (MLSI) represents fluctuations from the horizontal around the mediolateral axis The higher the value, the lower the mediolateral stability index.
Overall stability index (OASI) | 8 weeks
  The Biodex Balance System(Model 950-300, Biodex, Inc., Shirley, NY, USA) will be used to assess posture stability including overall stability index. It offers 12 levels of platform control and provides up to 20⁰ of surface tilt. Before the participant stepped onto the Biodex Balance System, the platform was in the "locked" position. Participants' data and test parameters were inserted. The parameters will be included trial time (20 seconds), number of trials (3 trials), and in between trials rest (10 seconds). Initial and end stability levels will be set from more to less stable (8-1) respectively. Overall stability index (OSI) is a composite of MLSI and APSI so it is sensitive to changes in both directions. These indices are standard deviations assessing fluctuations around the zero point from the horizontal rather than around the group mean. Higher values indicate more deviations and poor balance control
Pain intensity level | 8 weeks
  The visual analog scale (VAS) will be used to assess pain severity for all participants before and after the treatment. It is a valid pain rating scale and it is used to assess pain severity. It consists of a 10 cm straight line with two end points such as 0 is 'no pain at all' and 10 'pain as worse pain.
Pain pressure threshold (PPT) | 8 weeks
  The pressure algometry (12-0303 Push-Pull Force Gauge, Fabrication Enterprises, Inc., USA) with a probe size of 1.0 cm2 will be used to assess pain pressure threshold for all participants before and after the treatment..
  The pressure will be applied on the trigger points at 3 cm lateral to the spinous processes (L1-S5).The reading was expressed in Kg/cm2.
  During PPT measurement, assessor will place the circular probe perpendicular to the skin and press, the participant will be asked to say "stop" when feels pressure or discomfort. Four consecutive PPT measures will be performed at each site with 30 seconds of rest between measurements then the PPT of all trigger points will be averaged and used for analysis.

SECONDARY OUTCOMES:
Assessment of function disability | 8 weeks
  The Arabic version of Oswestry Disability Index (ODI) will be used to assess the function disability level of all participants before and after treatment. It consists of ten sections with six responses about daily activities. For each section the total score is 5; if the first statement is marked the score = 0; if the last statement is marked the score = 5. Intervening statements are scored according to rank. If more than one box is marked in each section, take the highest score. If all ten sections are completed the score is calculated as follows: Example: 16 (total score) of 50 (total possible score) × 100 = 32 %. If one section is missed (or not applicable) the score is calculated as follows: Example: 16 (total score)/45 (total possible score) × 100 = 35.6 %. A low score = low degree of disability, a high score = high degree of disability

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Awad, professor, Study Director — Cairo University; Dalia Kamel, Professor, Study Chair — Cairo University
Locations (1):
- Mohamed Khalaf Sayed, Cairo, Egypt